CLINICAL TRIAL: NCT00208871
Title: An Evaluation of Stereoscopic Digital Mammography for Earlier Detection of Breast Cancer and Reduced Rate of Recall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: BBN Technologies (Industry)
Responsible Party: Principal Investigator, Carl J. D'Orsi, MD, Proffessor of Radiology & Hematology/Oncology, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB00045816
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
Keywords: Stereoscopic digital mammography; Breast cancer detection; Reduced rate of recall; Focal abnormalities detection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Stereoscopic Digital Mammography — screening digital 3D mammogram

SUMMARY:
The primary goal of this study is to compare, within a clinical screening setting, the performance of stereoscopic digital mammography with standard (non-stereo) digital mammography in the detection of abnormalities in the breast, including early breast cancer.

DETAILED DESCRIPTION:
The clinical trial, begun in December, 2004, is being conducted at Emory University. Over the next three years, we will enroll and image about 2000 women who are at elevated risk for development of breast cancer (personal or family history of breast cancer) as they come in for their annual screening examinations. Each participating patient will be imaged with both systems, and the stereo and standard (non-stereo) images will be read independently by different mammographers.

A stereoscopic digital mammogram consists of two x-ray images of the breast acquired from slightly different points of view on a digital mammography unit. The x-ray source is rotated 10-degrees between the two exposures while the position of the breast remains fixed in the compression device. The stereo pair of mammograms is viewed on a new third-generation, high-resolution stereo display workstation that was developed in the first part of this project. The mammographer views the stereo display wearing lightweight polarized glasses, enabling him or her to see in depth the internal structure within the breast. As a result, a subtle lesion that may be obscured by superimposed normal tissue in a standard 2D image, now becomes visible as the overlying and underlying normal tissue is separated in depth. Conversely, layers of tissue that may falsely resemble a lesion in a standard 2D image due to chance superimposition, are seen in the stereo mammogram to lie at different depths and, thus, will not be mistaken as a lesion.

We anticipate that with stereo mammography the mammographers will detect subtle lesions in the stereo images that are missed in the non-stereo images. We also expect that there will be fewer false positive detections with the stereo images compared to the standard images. Finally, we also expect that the mammographers will be more confident in their judgments of what they see in the stereo images, resulting in a reduced rate of recall of patients for further work-up.

ELIGIBILITY:
Personal risk factors (any of the following)

* Personal history of breast and/or ovarian cancer, regardless of age.
* Prior breast biopsy that included any of the following high risk, benign lesion: Lobular carcinoma in-situ, Atypical ductal hyperplasia, Atypical lobular hyperplasia, Atypical columnar hyperplasia.
* Positive test for known mutations of BRCA 1 or 2 genes, regardless of age.
* History of chest irradiation for treatment of non-breast disease (EX:lymphoma, lung cancer) at least 15 years prior to enrollment.

Family history (over 30 years of age with any of the following, some exceptions may appy)

* Ashkenazi Jewish ancestry, regardless of age.
* Any history of male breast cancer on the maternal or paternal side.
* Breast and ovarian cancer in a close relative (mother, sister, daughter)
* Breast or ovarian cancer in more than one close relative (mother,sister daughter)
* Breast cancer in a close relative (mother, sister, daughter) with early onset(<50 years of age)
* Breast and ovarian cancer in a 2nd. degree relative (grandmother, aunt, niece) with early onset of breast cancer. (<50 years of age)
* Multiple history of breast cancer in 1st. and 2nd. degree relatives.

Exclusion Criteria:

* Patient does not meet any of the inclusion criteria,
* Patient has had breast augmentation, except for unilateral augmentation done for prior mastectomy,
* Patient has suspected or confirmed pregnancy,
* Patient has large breasts that cannot be adequately imaged on the 19 x 23 cm detector surface of the GE Senographe 2000D digital mammography unit.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1467 (Actual)
Dates: Start 2004-12; Primary Completion 2007-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
sensitivity/specificity | Aug '04 to Dec '07

SECONDARY OUTCOMES:
Recall rate | Aug '04 to December '7

CONTACTS AND LOCATIONS:
Overall Officials: David J Getty, Ph.D., Principal Investigator — BBN Technologies; Carl J D'Orsi, MD, Principal Investigator — Emory School of Medicine Site PI
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Getty DJ, Pickett RM, D'Orsi CJ. Stereoscopic digital mammography: improving detection and diagnosis of breast cancer. In: Computer Assisted Radiology and Surgery (CARS-2001). Berlin, Germany: Elsevier Science B.V., 2001.
- [Background] Getty D. J. Stereoscopic digital mammography. Proceedings of the First Americas Display Engineering and Applications Conference (ADEAC '04), Ft. Worth, 2004, 11-14.
- [Background] Getty, D. J. Stereoscopic and biplane digital radiography. In E. Samei & M. Flynn (Eds.), RSNA Categorical Course in Diagnostic Radiology Physics: Advances in Digital Radiography. RSNA Publications, 2003; 199-209.
- [Result] Getty, D. J. Stereoscopic digital mammography: perceptual and display factors leading to improved early detection of breast cancer. In H-O Peitgen (Ed.), Digital Mammography, IWDM 2002, 6th International Workshop on Digital Mammography. Berlin: Springer, 2003, 431-435.
- See also: clinical trials, stereoscopic digital mammography — http://www.cancer.emory.edu/